CLINICAL TRIAL: NCT01728298
Title: A Dose Response Evaluation of SLITone Ultra HDM Mix Immunotherapy - The SUMMIT Trial
Brief Title: A Dose Response Evaluation of SLITone Ultra HDM Mix Immunotherapy
Acronym: SUMMIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-M-01
Record Dates: First submitted 2012-11-02; First posted 2012-11-19 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Allergic Rhinitis
Keywords: House Dust Mite; allergy; rhinitis; asthma
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity; Rhinitis; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SLITone ULTRA low dose (Active Comparator): SLITone ULTRA HDM immunotherapy
  Interventions: Biological: SLITone ULTRA HDM immunotherapy
- SLITone ULTRA medium dose (Active Comparator): SLITone ULTRA HDM immunotherapy
  Interventions: Biological: SLITone ULTRA HDM immunotherapy
- SLITone ULTRA high dose (Active Comparator): SLITone ULTRA HDM immunotherapy
  Interventions: Biological: SLITone ULTRA HDM immunotherapy

INTERVENTIONS:
Biological: SLITone ULTRA HDM immunotherapy

SUMMARY:
The primary objective of the trial is to evaluate the dose-response relationship with regards to change in immunological parameters and safety for SLITone ULTRA house dust mite mix in adult subjects with moderate to severe HDM allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Moderate to severe persistent HDM allergic rhinitis with or without asthma
* Moderate to severe HDM allergic rhinitis symptoms during a baseline period
* Positive skin prick test response (wheal diameter ≥ 3 mm)
* Positive specific IgE ≥ IgE Class 2, ≥ 0.70 kU/l)

Exclusion Criteria:

* Previous treatment with immunotherapy with House dust mite immunotherapy
* Ongoing treatment with any allergen specific immunotherapy product
* Reduced lung function
* Clinical history of uncontrolled asthma
* Inflammatory conditions in the oral cavity with severe symptoms
* History of anaphylaxis with cardiorespiratory symptoms
* History of recurrent generalised urticaria
* A history of drug induced facial angioedema or hereditary angiooedema
* Any clinically relevant chronic disease (≥3 months duration)
* Systemic disease affecting the immune system
* Immunosuppressive treatment
* Currently treated with tricyclic antidepressants; catecholamine-Methyltransferase inhibitors and mono amine oxidase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in IgE-blocking factor after 6 months of treatment | 6 months

SECONDARY OUTCOMES:
Number of subjects with treatment related adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alain Didier, Pr., Principal Investigator — Hôpital Larrey, Toulouse
Locations (1):
- Proffesor Alain Didier, Toulouse, France